CLINICAL TRIAL: NCT01006343
Title: Dietary Pork, Appetite and Weight Loss in Human
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Wayne Campbell, Professor, Foods and Nutrition, Purdue University
Allocation: Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: 0504001915
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2009-10

CONDITIONS: Appetite; Weight Loss
MeSH Terms: conditions — Weight Loss

ARMS (2):
- Higher Protein (HP) (Experimental): Subjects will be required to follow their seven day menu plan for the 12 weeks of intervention. The HP menus will contain 30% protein, 45% carbohydrate, and 25% fat. Subjects in the HP group will be provided with portioned, cooked and frozen pork products as part of their HP menu plan.
  Interventions: Other: Higher Protein (HP)
- Lower Protein (LP) (Experimental): Subjects will be required to follow their seven day menu plan for the 12 weeks of intervention. The LP group menus will contain 18% protein, 57% carbohydrate, 25% fat. The LP group will follow a lacto-ovo vegetarian menu with no striated tissue foods. Subjects in the LP group will be provided with selected, portioned dairy products.
  Interventions: Other: Lower Protein (LP)

INTERVENTIONS:
Other: Higher Protein (HP)
  Arms: Higher Protein (HP)
Other: Lower Protein (LP)
  Arms: Lower Protein (LP)

SUMMARY:
The entire study protocol will last 13 weeks. Women will be randomly assigned to one of two experimental groups: high and low protein. All women will consume their unrestricted habitual diet during week 1 while baseline testing and measurements are taken. Starting at week 2, women in both groups will be counseled to consume a 750 kcal/day energy deficit diet containing either the RDA (LP group) or more than the recommended dietary allowance (RDA) (HP group) for protein. The energy restriction period will continue for 12 weeks (through study week 13) and is expected to result in body weight reduction of approximately 17 pounds. Testing and measurements will be repeated during week 13.

ELIGIBILITY:
Inclusion Criteria:

* Eligible women will have a body mass index (BMI: weight (kg)/height (m2)) ranging from 26-36.
* Must be at least 21 years old.

Exclusion Criteria:

* Women with medical conditions that might place them at risk for participating in the study or interfere with the successful completion of the study protocol will be excluded.
* BMI <26 or >36.
* Younger than 21 years old.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Purdue University, West Lafayette, Indiana, United States